CLINICAL TRIAL: NCT01843231
Title: A Randomized Controlled Multicenter Feasibility Study of an IncisionLEss Operating Platform for Primary ObeSiTy vs. Diet-exercise Alone: The MILEPOST Study
Brief Title: Use of the Incisionless Operating Platform as a Primary Treatment for Obesity vs. Diet-Exercise Alone
Acronym: MILEPOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 41936
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: g-Cath EZ Suture Anchor Delivery Catheter; Weight Loss Intervention
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- g-Cath EZ Treatment Group (Experimental): Evaluate the safety and effectiveness of the g-CathTM EZ Suture Anchor Delivery Catheter as an early weight loss intervention
  Interventions: Device: g-CathTM EZ Suture Anchor Delivery Catheter
- Diet and exercise Control Group (Active Comparator): Diet and Exercise only control group
  Interventions: Other: Diet and Exercise Control Group

INTERVENTIONS:
Device: g-CathTM EZ Suture Anchor Delivery Catheter — Use of the g-Cath EZ Suture Anchor Delivery Catheter for the placement of g-cath EZ suture anchors as an early weight loss intervention + diet and exercise as compared to those in the diet and exercise control group
  Arms: g-Cath EZ Treatment Group
Other: Diet and Exercise Control Group — Patients in a diet and exercise only control group that will be compared to those in the g-Cath EZ Suture Anchor Delivery Catheter treatment group
  Arms: Diet and exercise Control Group

SUMMARY:
This study is a multi-center, open/unblended study (3:1Treatment: Control) to evaluate the safety and effectiveness of the g-Cath EZ Suture Anchor Delivery Catheter as an early weight loss intervention compared to a diet and exercise control only. Mean % Total Body Weight Loss [TBWL] in Treatment subjects versus that of Control subjects at 12 months is the primary endpoint. The proportion of subjects achieving ≥ 5% TBWL at 12 months in the treatment group is a co-primary endpoint.

DETAILED DESCRIPTION:
This study will evaluate the safety and effectiveness of the g-Cath EZ Suture Anchor Delivery Catheter as an early weight loss intervention compared to a diet and exercise control only. The weight loss outcomes will be used to assess treatment effect. This study is a multi-center, open/unblinded, prospective randomized feasibility study (3:1Treatment: Control) study. Patients in the control group will be offered the opportunity to crossover to the treatment group at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* Body Mass Index [BMI] of >30 and <40 with or without a co-morbid condition
* Subject has failed more conservative weight reduction alternatives such as supervised diet, exercise or behavior modification programs in the last year
* No significant weight change (+/- 5% of total body weight) in last 6 months
* American Society Anesthesiologists-Physical Status score ≤ 2 (Appendix III),
* Subject agrees not to have any additional weight loss interventional procedures or liposuction for at least 30 months following study enrollment,
* Has not taken any prescription or over the counter weight loss medications for at least 6 months,
* Signed informed consent.
* Subject is willing to cooperate with post-operative dietary recommendations and assessment tests,

Exclusion Criteria:

* History of (or intraoperative evidence of) bariatric, gastric or esophageal surgery
* Esophageal stricture or other anatomy and/or condition that could preclude passage of endolumenal instruments
* Severe gastroesophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with prescription drug therapy
* Known hiatal hernia >3 centimeters by history or as determined by Upper Gastrointestinal exam or endoscopy
* Pancreatic insufficiency/disease
* Active peptic ulcer
* Pregnancy or plans of pregnancy in the next 12 months
* Present Corticosteroid Use
* History of inflammatory disease of Gastrointestinal [GI] tract; Coagulation disorders; hepatic insufficiency or cirrhosis
* History or present use of insulin or insulin derivatives for treatment of diabetes
* Type II Diabetes Mellitus [DM] (as defined by Glycosylated Hemoglobin [HgbA1c] >6.5) for greater than 2 years at the time of enrollment
* Uncontrolled Type II DM (HgbA1c > 7.0 at screening)
* Quit smoking within last 6 months at time of enrollment or plans to quit smoking in the next year
* Immunosuppression
* Portal hypertension and/or varices
* Active gastric ulcer disease
* Gastric outlet obstruction or stenosis
* Beck Depression Inventory (Short) Score ≥12 (see Appendix IV);
* Subject has a history of drug or alcohol abuse or actively abusing either as defined by Cage and DAST [drug use] questionnaires or positive Urinalysis [UA] drug screen
* Severe disturbances in eating behavior (i.e. binge eating)
* Known presence of a significant depression, psychosis, or other mood or eating disorder
* Actively treated depression (except for stable treated depression for >1year and normal [Beck Depression Inventory [BDI] and psych exam)
* Present or past history of psychosis or other mood or eating disorder
* Non-ambulatory or has significant impairment of mobility
* Known hormonal or genetic cause for obesity with the exception of treated hypothyroidism.
* Participating in another clinical study
* Is a first degree relative of investigator, or support staff involved in the study.
* Employed by investigator or institution involved in the study
* Subject is not able to provide written informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 12 months
  Incidence and severity of Adverse Events [AE] over 12 Months
Primary Efficacy Endpoint | 12 months
  Mean % TBWL at 12 months for Treatment subjects compared to Control subjects
Co-Primary Efficacy Endpoint | 12 months
  The proportion of Treatment subjects achieving ≥ 5% TBWL at 12 months

SECONDARY OUTCOMES:
First Secondary Efficacy Endpoint | 24 months
  Mean % TBWL at 24 months.
Second Secondary Efficacy endpoint | 24 months
  Proportion of subjects achieving ≥ 5% TBWL at 24 months
Third Secondary Efficacy endpoint | 2, 6, 12 months
  Satiety changes (volume and time to satiety at 2, 6, 12 months post-procedure)
Fourth Secondary Efficacy endpoint | 12 & 18 months
  % Estimated Weight Loss [EWL] at 12 months and 18 months [% EWL will be calculated using BMI-25 criteria]

CONTACTS AND LOCATIONS:
Overall Officials: Jorge C. Espinos, Dr., Principal Investigator — Centro Medico Teknon
Locations (3):
- Krakenhaus Hallein, Hallein, Salzburg, Austria
- Atrium Medical Centre, Heerlen, Netherlands
- Centro Medico Teknon, Barcelona, Spain

REFERENCES:
- [Derived] Miller K, Turro R, Greve JW, Bakker CM, Buchwald JN, Espinos JC. MILEPOST Multicenter Randomized Controlled Trial: 12-Month Weight Loss and Satiety Outcomes After pose SM vs. Medical Therapy. Obes Surg. 2017 Feb;27(2):310-322. doi: 10.1007/s11695-016-2295-9. PMID 27468907